CLINICAL TRIAL: NCT05676762
Title: Le Conseil Minimal Autour de la Contraception : Quel Impact Sur la Prise de Conscience du Risque de Grossesse Non désirée et Sur l'Attrait à la Contraception
Brief Title: Contraceptive Counselling: Impact on Awareness of the Risk of Unwanted Pregnancy and on the Appeal of Contraception
Acronym: CMC
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Centre Hospitalier Universitaire de la Réunion (Other)
Responsible Party: Sponsor
Other Study IDs: 2021/CHU/34
Record Dates: First submitted 2022-07-21; First posted 2023-01-09 (Actual); Last update posted 2023-01-09 (Actual); Status verified 2022-07

CONDITIONS: Contraception

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The hypothesis of this study is that the generalisation of minimal contraceptive advice in general medical consultations among women of childbearing age in Reunion Island who do not use contraception but who have sexual relations and do not wish to become pregnant within the year could induce an awareness of the risk of unwanted pregnancy and lead to a change in behaviour with regard to contraceptive methods.

ELIGIBILITY:
Inclusion Criteria:

* Women from 18 to 50 years old
* Consulting in a general practice in Reunion Island
* French or Creole speaking
* Not having any contraceptive means
* Having sexual intercourse
* Not having any desire to become pregnant within the year
* Collection of non-opposition

Exclusion Criteria:

* Consultation for a desire or follow-up of a pregnancy
* Consultation for an abortion
* Consultation for a contraceptive method
* Known infertility
* Inability to answer the telephone (hearing impaired, mute)
* Severe cognitive disorder (mental retardation, dementia, active psychosis)
* Women under guardianship or curatorship

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: On the basis of 30 participating GPs, the estimation of the number of inclusions is 400 women, which seems sufficient for this study.
  The desired number of inclusions is 45 women/month (400 women over 9 months).
Sampling Method: Non-Probability Sample
Enrollment: 117 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2023-01-15 (Estimated)

PRIMARY OUTCOMES:
Impact of a minimal councelling regarding the contraception awareness of risk of unwanted pregnancy | between Day 1 and Month 1
  Change of Proportion of women with no contraception and having sexual relations without a desire of pregnancy

CONTACTS AND LOCATIONS:
Overall Officials: Sébastien LERUSTE, MD, Principal Investigator — Universite de La Reunion
Locations (1):
- Cabinet de médecine générale, Saint-Philippe, Reunion

IPD SHARING:
Plan to Share IPD: No